CLINICAL TRIAL: NCT01800708
Title: The Use of Intraocular Triamcinolone in the Perioperative Period of Congenital Cataract Surgery
Brief Title: Cataract Surgery With Intracameral Triamcinolone in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundação Altino Ventura (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2013-02-25; First posted 2013-02-28 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triamcinolone acetonide (Active Comparator): The study group will receive an intraoperative intracameral injection of triamcinolone acetonide
  Interventions: Drug: Triamcinolone acetonide
- Prednisolone syrup (Active Comparator): The control group will receive prednisolone syrup postoperatively
  Interventions: Drug: Prednisolone syrup

INTERVENTIONS:
Drug: Triamcinolone acetonide
  Other Names: Triancinolona Ophthalmos
  Arms: Triamcinolone acetonide
Drug: Prednisolone syrup
  Arms: Prednisolone syrup

SUMMARY:
The aim of the present study is to investigate the outcomes of congenital cataract surgery when injecting intraoperative intracameral triamcinolone versus the postoperative use of oral prednisolone.

This is a prospective, randomized clinical trial. Sixty children will be submitted to congenital cataract surgery younger than 2 years of age. They will be randomly divided in two groups. The study group will receive an intraoperative intracameral triamcinolone acetonide injection. The control group will receive prednisolone syrup postoperatively. The surgical outcomes will be assessed after one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients younger than 2 years of age
* Unilateral or bilateral congenital cataracts compromising the red reflex

Exclusion Criteria:

* Corneal opacity
* Glaucoma
* Aniridia
* Subluxated cataract
* Traumatic cataract
* Complex microphthalmia
* Persistant hyperplastic primary vitreous
* Retinal detachment
* Patients with intraoperative complications, such as IOL implanted in the sulcus

Ages: 6 Weeks to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Visual axis obscuration | 1 year after surgery
  Visual axis obscuration will be evaluated under sedation, with a dilated pupil. All patients will be classified by the principal investigator as having or not a significant visual axis obscuration, based on the red reflex.
Intraocular pressure | 1 year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Ventura, MD, Principal Investigator — Fundação Altino Ventura
Locations (1):
- Altino Ventura Foundation, Recife, Pernambuco, Brazil